#### **PARTICIPANT CONSENT FORM**

Study title: Personal and environmental correlates of problematic internet and smartphone use

**Principal investigator:** Yumei LI **Document data:** June 6, 2022

About this project

My name is Yumei LI. I am a PhD student at the City University of Hong Kong working with my supervisor, Dr. KWOK LAI Yuk Ching Sylvia, in the School/ Department of Social & Behavioural Sciences. We would like to invite you to participate in our problematic technology use intervention program, which is designed to help participants reduce problematic internet and smartphone use behaviors through cognitive behavioral intervention techniques. The College Human Subjects Ethics Sub-Committee, College of Liberal Arts and Social Sciences has approved the project. Whether to participate in our intervention is entirely up to your personal decision.

# Study procedure

We will invite you to participate in an intervention program (four-week, 1 session per week, 90 minutes per session). Before the intervention, we refined our intervention design by conducting in-depth interviews with 30 participants. The current intervention involves the identification of character strengths (the first week), the perception of the meaning of life (the second week), the learning of strategies to develop hope (the third week), and the learning of emotion regulation strategies (the fourth week). At the beginning of the intervention, we will invite you (and the guardians of children under the age of 18) to sign the Informed Consent Form for Study. If you do not wish to do so, you may decline the invitation and withdraw from the study at any time. A professional social worker will guide all parts of the intervention.

#### Possible risks and discomfort

Our intervention will not bring you any physical or mental harm. Participating in this project will take up your 90 minutes per week over four weeks.

#### Participating in the study may bring you or society benefits

We hope that this intervention program will help reduce your risk of developing problematic Internet and smartphone use behaviors and enhance your positive development. In addition, the results of the intervention will help construct an intervention guidebook to guide future intervention activities for problematic Internet and smartphone use in at-risk populations.

### **Declaration of confidentiality**

This intervention project requires the collection of your name and contact information for the sole purpose of matching your personal data in the overall intervention process. We will do our best to ensure the confidentiality of your information. Except for the members of the research team, no one can associate your name with your participation, and it is impossible to know your answer to any specific question. The information you provide will only be used for research. The study data will be stored in a dedicated computer file. We will set a password for all computer files and store the computer in a locked office. Only the staff of this study can access these materials.

### Voluntary participation and withdrawal

Your participation is entirely **voluntary**. You will not receive any compensation or payment in return for your participation. At any stage, if you do not want to answer questions or continue to participate, you can stop the study and withdraw from the intervention without any adverse consequences.

#### Participant's rights

All projects involving human participation will be reviewed by the ethics committee to protect your rights and interests. If you have any questions, comments or concerns about research participation or the research itself, please feel free to contact the research investigator Yumei LI (PhD student of the Department of Social and Behavioural Sciences, City University of Hong Kong). Contact: +852 64078719 or +86 15527160797 or <a href="https://livensets.org/livensets/livens

### **Reply Slip-Participants**

# Project title: Personal and environmental correlates of problematic internet and smartphone use

If you agree to take part in the research, please sign your name below. Signing your name means you are agreeing that:

- (1) You have read and understood the Participant Information Sheet,
- (2) Questions about your participation in this study have been answered satisfactorily,
- (3) You are aware of the potential risks (if any), and
- (4) You are taking part in this research study voluntarily (without coercion).

| Printed Name of Participant: |
|------------------------------|
| Signature of Participant: |
| Date: |

# **Reply Slip-Guardians (For children under 18)**

# Project title: Personal and environmental correlates of problematic internet and smartphone use

If you agree your children to take part in the research, please sign your name below. Signing your name means you are agreeing that:

- (1) You have read and understood the Participant Information Sheet,
- (2) Questions about your child's participation in this study have been answered satisfactorily,
- (3) You are aware of the potential risks (if any), and
- (4) Your child is taking part in this research study voluntarily (without coercion).

| Printed Name of Child: |
|-------------------------------|
| Printed Parent/Guardian Name: |
| Signature of Parent/Guardian: |
| Date: |